CLINICAL TRIAL: NCT03505775
Title: Evaluation of the Muscular and Cutaneous Sodium Storage by 23Na Magnetic Resonance Imaging in Patients With Chronic Adrenal Insufficiency Compared to Healthy Subjects
Brief Title: Evaluation of the Muscular and Cutaneous Sodium Storage by 23Na MRI in Patients With Chronic Adrenal Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23NaMRT-AI
Record Dates: First submitted 2018-04-12; First posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Adrenal Insufficiency
Keywords: Hormone replacement; Mineralocorticoids; 23Na-magnetic resonance imaging; Tissue sodium content
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 23Na-MRI (Other): A 23Na magnetic resonance imaging of the calf (muscle and skin) was performed in every participating patient after clinical and laboratory examinations.
  Interventions: Diagnostic Test: 23Na magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: 23Na magnetic resonance imaging — Imaging/diagnostic: Evaluation of the muscular and cutaneous sodium storage by 23Na magnetic resonance imaging. 23Na magnetic resonance imaging: 23NA-MRI protocol on a 3T scanner (Magnetom PRISMA, Siemens, Erlangen) implementing a 3D sequence.

SUMMARY:
This study investigates the sodium content in the calf muscle and the skin obtained via 23Na-magnetic resonance imaging in patients with chronic adrenal insufficiency compared to healthy controls.

DETAILED DESCRIPTION:
Patients with chronic adrenal insufficiency depend on lifelong glucocorticoid and mineralocorticoid replacement therapy. Monitoring is based on clinical and laboratory parameters reflecting hemodynamic stability, electrolyte status and plasma renin concentration. Reduced subjective well-being is however often described by these patients in absence of clinical or laboratory abnormalities and is thus a strong indicator of the gap between the concept of adequate hormone substitution and patients' requirements. This study investigates the sodium content in the calf muscle and the skin obtained via 23Na-magnetic resonance imaging (MRI) in patients with chronic adrenal insufficiency compared to age-, sex- and BMI- matched healthy controls. The aim of the study is to evaluate the potential role of 23Na-MRI for monitoring of hormone replacement by investigating tissue sodium concentrations in patients with adrenal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Written informed consent
* Chronic adrenal insufficiency (first diagnosis > 6months), stable hormone replacement therapy with glucocorticoids (no dose-adjustment >50mg hydrocortisone within the last 8 weeks) and mineralocorticoids (only primary adrenal insufficiency)! Or healthy control (no adrenal insufficiency, normal serum-electrolytes, normotensive blood pressure, no medication with a known influence on the electrolyte balance)!

Exclusion Criteria:

* Pregnancy or breast-feeding
* Metal-implant (not MRI-compatible)
* Claustrophobia
* Chronic internistic disease (hypertension, heart failure, liver cirrhosis)
* Polydipsia (>4l/d)
* Long-term medication that can cause a hyponatraemia (for example diuretics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Muscle sodium content | 6 months
  Assessment of the sodium content of the calf muscle. Relative sodium signal intensities were calculated as ratio of tissue sodium intensity and the intensity of a vial containing a concentration of 100mmol/l.
Skin sodium content | 6 months
  Assessment of the sodium content of the calf skin. Relative sodium signal intensities were calculated as ratio of tissue sodium intensity and the intensity of a vial containing a concentration of 100mmol/l.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Hahner, MD, Prof., Principal Investigator — University Hospital Wuerzburg, Dept. of medicine I, Germany
Locations (1):
- University Hospital Wuerzburg, Dept. of medicine I, Würzburg, Germany

REFERENCES:
- [Background] Hahner S, Loeffler M, Fassnacht M, Weismann D, Koschker AC, Quinkler M, Decker O, Arlt W, Allolio B. Impaired subjective health status in 256 patients with adrenal insufficiency on standard therapy based on cross-sectional analysis. J Clin Endocrinol Metab. 2007 Oct;92(10):3912-22. doi: 10.1210/jc.2007-0685. Epub 2007 Aug 7. PMID 17684047
- [Background] Quinkler M, Oelkers W, Remde H, Allolio B. Mineralocorticoid substitution and monitoring in primary adrenal insufficiency. Best Pract Res Clin Endocrinol Metab. 2015 Jan;29(1):17-24. doi: 10.1016/j.beem.2014.08.008. Epub 2014 Aug 27. PMID 25617169
- [Background] Kopp C, Linz P, Dahlmann A, Hammon M, Jantsch J, Muller DN, Schmieder RE, Cavallaro A, Eckardt KU, Uder M, Luft FC, Titze J. 23Na magnetic resonance imaging-determined tissue sodium in healthy subjects and hypertensive patients. Hypertension. 2013 Mar;61(3):635-40. doi: 10.1161/HYPERTENSIONAHA.111.00566. Epub 2013 Jan 21. PMID 23339169
- [Background] Kopp C, Linz P, Wachsmuth L, Dahlmann A, Horbach T, Schofl C, Renz W, Santoro D, Niendorf T, Muller DN, Neininger M, Cavallaro A, Eckardt KU, Schmieder RE, Luft FC, Uder M, Titze J. (23)Na magnetic resonance imaging of tissue sodium. Hypertension. 2012 Jan;59(1):167-72. doi: 10.1161/HYPERTENSIONAHA.111.183517. Epub 2011 Dec 5. PMID 22146510